CLINICAL TRIAL: NCT02209103
Title: Determination of the Sleep Improving Effects of Phenolics From an Orange Peel Extract
Brief Title: The Sleep Improving Effects of Orange Phenolics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NL43845.068.13
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2014-08

CONDITIONS: Polyphenols; Sleep; Fatigue
Keywords: Polyphenols; Orange; Sleep; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Citrus flavonoid (Experimental): Citrus flavonoid
  Interventions: Dietary Supplement: Lozenge containing citrus flavonoid
- Citrus flavonoid formulation (Experimental): Citrus flavonoid formulation
  Interventions: Dietary Supplement: Lozenge containing citrus flavonoid formulation
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Identical looking placebo

INTERVENTIONS:
Dietary Supplement: Lozenge containing citrus flavonoid
  Arms: Citrus flavonoid
Dietary Supplement: Lozenge containing citrus flavonoid formulation
  Arms: Citrus flavonoid formulation
Dietary Supplement: Identical looking placebo
  Arms: Placebo

SUMMARY:
This study aims to determine whether a citrus flavonoid or a citrus flavonoid formulation can improve objective sleep duration and/or quality, and/or improve perceived sleep quality and feelings of rest.

Participants will complete a total of 9 test nights, which consist of sleeping with the sleep monitoring system after ingestion of the test product or a placebo, and filling out sleep-related questionnaires.

The study has a crossover design, meaning that all participants receive all three interventions (citrus flavonoid, citrus flavonoid formulation, placebo) three times, in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Non-smoking
* Healthy
* Lightly disturbed sleep for at least six months, on a regular basis

Exclusion Criteria:

* Severe sleep disorders (sleep apnea, restless legs syndrome)
* An apparent cause for the sleep disorders (pain, etc.)
* Clinically significant abnormal liver functioning
* Clinically significant abnormal serum creatinine
* BMI lower than 18 or higher than 30 kg/m2
* Use of concomitant medications or supplements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Sleep quality as assessed objectively by means of a portable sleep monitoring system (ZEO) | 9 test nights (up to 9 days)
  • The primary endpoint for this study is the determination of sleep quality, as assessed objectively with the portable sleep monitoring system ZEO, which is based on EEG/EMG (electromyography) coupled with an automatic sleep phase classifier. Sleep stages are classified as deep sleep, light sleep, REM (rapid eye movement) sleep or awake. The sleep patterns of the participants after ingestion of the two different test products will be compared to each other and to placebo.

SECONDARY OUTCOMES:
Subjective sleep quality ratings and fitness, tiredness and cognitive ratings, obtained from questionnaires | up to 9 days. Questionnaires are filled out the morning after every test night
  Leeds Sleep Evaluation Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chris Van der Grinten, Principal Investigator — Department: lung diseases MUMC
Locations (1):
- Maastricht University Medical Center (MUMC), Maastricht, Netherlands